CLINICAL TRIAL: NCT00612794
Title: Multiple-Dose Study to Examine Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY2148568 Long-Acting Release in Japanese Patients With Type 2 Diabetes Mellitus
Brief Title: A Study to Examine Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Exenatide Once Weekly in Japanese Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H8O-JE-GWBW
Record Dates: First submitted 2008-01-30; First posted 2008-02-12 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-01

CONDITIONS: Type 2 Diabetes
Keywords: exenatide; Byetta; diabetes; Amylin; Lilly
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): exenatide once weekly, 0.8mg
  Interventions: Drug: exenatide once weekly
- 2 (Experimental): exenatide once weekly, 2.0mg
  Interventions: Drug: exenatide once weekly
- 3 (Placebo Comparator): volume equivalent to 0.8mg of exenatide once weekly
  Interventions: Drug: placebo
- 4 (Placebo Comparator): volume equivalent to 2.0mg of exenatide once weekly
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: exenatide once weekly — subcutaneous injection, once weekly
  Arms: 1; 2
Drug: placebo — subcutaneous injection, once weekly
  Arms: 3; 4

SUMMARY:
Exenatide twice daily has been studied in Japanese type 2 diabetes patients. A once-weekly version of exenatide is currently being evaluated. Study GWBW is the first study of exenatide once weekly in Japanese patients. This study is designed to evaluate safety and tolerability of exenatide once weekly in Japanese patients and determine whether the dose selected for US and European development is appropriate for Japanese patients with Type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Body weight ≥50 kg.
* Have suboptimal glycemic control as evidenced by an HbA1c defined by the following criteria: *6.5% to 10.0%, inclusive, at study start for patients managed with diet modification and exercise or treated with oral antidiabetics drug but not alpha glucosidase inhibitor or meglitinide derivatives; *6.5% to 9.5%, inclusive, at study start for patients treated with oral antidiabetics including alpha glucosidase inhibitor or meglitinide derivatives.
* Have been treated with diet modification and exercise alone or in combination with a stable regimen of oral antidiabetic drugs (sulfonylurea, metformin and thiazolidinedione) for at least 2 months prior to study start. In the case of patients with concomitant use of sulfonylurea, the dose of sulfonylurea must not be more than maximum recommended dose. The patients with concomitant use of alpha glucosidase inhibitors (Glucobay® [acarbose], Basen® [voglibose], or Seibule® [miglitol]) or meglitinide derivatives (Glufast® [mitiglinide] or Fastic®/Starsis® [nateglinide]) can be included in this study, but these drugs must be discontinued after confirmation of eligibility at study start.

Exclusion Criteria:

* Subjects who have donated more than 200 mL of blood and component blood donation within one month of study start, or those who have donated more than 400 mL of blood within three months of study start.
* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.
* Have participated and received at least one dose of exenatide or other GLP-1 analogs in this study previously, or any other study using exenatide or other GLP-1 analogs.
* Are treated with any exogenous insulin within 3 months of screening.
* Are continuously treated with any of the following excluded medications within 3 months of screening (more than 7 days per 1 month): *Drugs that directly affect gastrointestinal motility, including Nauzelin® (domperidone), Primperan®/Terperan® (metoclopramide), Ganaton® (itopride), Acenalin® (cisapride), Gasmotin® (mosapride), or Cerekinon® (trimebutine).
* Females who are breastfeeding.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-09; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of exenatide administered once weekly by subcutaneous (SC) injection in subjects with type 2 diabetes mellitus. | 10 weeks

SECONDARY OUTCOMES:
To assess the pharmacokinetics of exenatide administered once weekly by SC injection in subjects with type 2 diabetes mellitus. | 10 weeks
To explore the pharmacodynamics of exenatide administered once weekly by SC injection in subjects with type 2 diabetes mellitus regarding the following: *fasting and postprandial glucose concentrations; *HbA1c; *Body weight. | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, MD, Study Director — Eli Lilly and Company
Locations (4):
- Japan (4):
  - Research Site, Fukuoka
  - Research Site, Kanagawa
  - Research Site, Osaka
  - Research Site, Tokyo

REFERENCES:
- [Derived] Iwamoto K, Nasu R, Yamamura A, Kothare PA, Mace K, Wolka AM, Linnebjerg H. Safety, tolerability, pharmacokinetics, and pharmacodynamics of exenatide once weekly in Japanese patients with type 2 diabetes. Endocr J. 2009;56(8):951-62. doi: 10.1507/endocrj.k09e-147. Epub 2009 Aug 25. PMID 19706990